CLINICAL TRIAL: NCT02172248
Title: Relative Bioavailability of Both BI 10773 and Metformin After Coadministration Compared to Multiple Oral Doses of BI 10773 (50 mg q.d.) Alone and Metformin (1000 mg b.i.d.) Alone to Healthy Male Volunteers (an Open-label, Randomised, Crossover, Clinical Phase I Study)
Brief Title: Relative Bioavailability BI 10773 and Metformin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.6
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

ARMS (2):
- Sequence ABC (Experimental): 1. Treatment A: BI 10773 once daily from day 1 to 5
  2. Treatment B: BI 10773 once daily from day 1 to 4 and metformin twice daily from day 1 to 3 and once in the morning on day 4
  3. Treatment C: metformin twice daily from day 1 to 3 and once in the morning on day 4
  Interventions: Drug: BI 10773; Drug: Metformin
- Sequence CAB (Experimental): 1. Treatment C: metformin twice daily from day 1 to 3 and once in the morning on day 4
  2. Treatment A: BI 10773 once daily from day 1 to 5
  3. Treatment B: BI 10773 once daily from day 1 to 4 and metformin twice daily from day 1 to 3 and once in the morning on day 4
  Interventions: Drug: BI 10773; Drug: Metformin

INTERVENTIONS:
Drug: BI 10773
Drug: Metformin

SUMMARY:
The objective was to investigate a possible drug-drug interaction between BI 10773 and metformin when co-administered as multiple oral doses. Therefore, the relative bioavailabilities of BI 10773 and metformin were determined when both drugs were given in combination compared with BI 10773 or metformin given alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP (Blood Pressure), PR (Pulse Rate)), 12-lead ECG (Electrocardiogram), clinical laboratory tests
* Age 18 to 50 years (incl.)
* BMI (Body Mass Index) 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 30 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 7 days
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 7 days

SECONDARY OUTCOMES:
C24,N (concentration of analyte in plasma at 24 hours post-drug administration after administration of the Nth dose) of BI 10773 | up to 7 days
C12,N (concentration of analyte in plasma at 12 hours post-drug administration after administration of the Nth dose) of metformin | up to 7 days
λz,ss (terminal half-life of the analyte in plasma) | up to 7 days
t½,ss (terminal half-life of the analyte in plasma at steady state) | up to 7 days
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 7 days
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 7 days
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | up to 7 days
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 7 days
Aet1-t2,ss (amount of analyte eliminated in urine at steady state over a uniform dosing interval τ) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
fet1-t2,ss (fraction of analyte excreted unchanged in urine at steady state over a uniform dosing interval τ) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
CLR,ss (renal clearance of the analyte at steady state) of BI 10773 and metformin | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
Urinary glucose excretion (UGE) | 1 hour pre-dose, 0-2, 2-4, 4-8, 8-12, 12-24 hours after last dosing
Number of patients with abnormal findings in physical examination | Baseline and within 3-14 days after last study drug administration
Number of patients with clinically significant changes in vital signs (Blood Pressure, Pulse Rate) | Baseline, day 1 and within 3-14 days after last study drug administration
Number of patients with abnormal findings in 12-lead ECG (electrocardiogram) | Baseline and within 3-14 days after last study drug administration
Number of patients with abnormal changes in clinical laboratory tests | Baseline, day 1, 4, 5 and within 3-14 days after last study drug administration
Number of patients with adverse events | up to 40 days
Assessment of tolerability by investigator on a 4-point scale | Within 3-14 days after last study drug administration